CLINICAL TRIAL: NCT04612309
Title: Retrospective Observational Study on the Use of Immunotherapy With Anti PD-1 Antibodies in Patients With MSI-H Metastatic Colorectal Cancer
Brief Title: Retrospective Study on the Use of Immunotherapy in Patients With MSI-H Metastatic Colorectal Cancer
Acronym: C-MSI
Status: Active, not recruiting | Type: Observational
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Responsible Party: Sponsor
Other Study IDs: GOIRC-07-2019
Record Dates: First submitted 2020-09-30; First posted 2020-11-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer
Keywords: H-MSI; immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treated: Patient with colorectal cancer already treated with immunotherapy
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Drug: Immunotherapy — patient treated with at least 1 immunotherapy administration

SUMMARY:
An increasing number of patients with metastatic colorectal cancer (mCRC) are able to receive 3 or more lines of therapy. In this setting, can be recognize treatments such as regorafenib (an oral multikinase inhibitor), trifluridine/tipiracil hydrochloride (TAS-102), an antineoplastic nucleoside analogue, and antibodies anti-epidermal growth factor receptor (EGFR) in patients with RAS wild-type tumors (if no prior exposure to antibodies). Maintaining quality of life is an essential goal for third- and later-line treatments for patients.

The anti-programmed cell death protein 1 (anti-PD-1) immune checkpoint inhibitors, pembrolizumab and nivolumab, were approved in the US by the FDA in 2017, and the combination nivolumab plus ipilimumab (anti CTLA-4) was recently approved by the FDA in 2018, all in the second and later-line setting for patients with microsatellite instability-high (MSI-H) or deficient DNA mismatch repair mCRC whose disease has progressed despite treatment with fluoropyrimidine-, oxaliplatin-, and irinotecan-based chemotherapy. At present, these agents are not approved in Europe for mCRC patients with MSI-H. Clinical trial results and scientific data supported evidence that immunotherapies provide benefit but are limited to the small proportion (< 5%) of patients with MSI-H tumors, in whom they are highly effective. Therefore, patients with MSI-H disease should be referred as expeditiously as possible to receive immune checkpoint inhibitors.

The aim the study is to retrospectively collect data of patients treated with immunotherapy in the context of real clinical practice, in order to describe the real impact in terms of clinical outcomes and tolerability of treatment in common clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent for alive patients
* Patients with diagnosis of colorectal cancer with MSI-H
* Patient treated with at least one administration of antibody anti PD-1 for colorectal cancer prior to 30 June 2020 outside clinical trials.
* Availability of the tumor tissue from the primary tumor or a metastatic site for molecular analyses. The availability of tumor tissue is recommended but not mandatory.

Exclusion Criteria:

* Patients who received immunotherapy during a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer treated with at least one administration of immunotherapy prior to 30 June 2020
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
effectiveness | 6 months after the start of immunotherapy
  survival rate of patients

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Pinto, MD, Study Chair — Gruppo Oncologico Italiano di Ricerca Clinica
Locations (1):
- Ospedale Ramazzini, Carpi, Modena, Italy

IPD SHARING:
Plan to Share IPD: Yes